CLINICAL TRIAL: NCT02412605
Title: Effect of Trophectoderm Biopsy for Sex Selection on the Pregnancy and Miscarriage Rates of Women Undergoing IVF/ICSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Other Study IDs: PGD2
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Assisted Reproduction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fertile embryo biopsy: Fertile couples requesting sex selection for family balancing
  Interventions: Procedure: Trophectoderm embryo biopsy
- Infertile embryo biopsy: Infertile women having embryo biopsy
  Interventions: Procedure: Trophectoderm embryo biopsy
- IVF/ICSI: Infertile women undergoing IVF/ICSI without embryo biopsy

INTERVENTIONS:
Procedure: Trophectoderm embryo biopsy — Day 5 embryos were incubated in calcium/Magnesium free culture. A laser beam was used to produce a hole in the zona pellucida. Trophectoderm cells were collected by gentle suction using the biopsy pipette.
  Florescent in situ hybridization of the trophectoderm nuclei with probes specific to the X- and Y-chromosomes was performed. the embryos were frozen and the cycles deferred.The embryos were thawed in the following cycle and if possible 2 embryos of the desired sex were transferred.
  Groups: Fertile embryo biopsy; Infertile embryo biopsy

SUMMARY:
Records of women who had trophectoderm biopsy for sex selection over the last 3 years will be reviewed and its outcome will be compared to other records of women who had IVF/ICSI without embryo biopsy.

DETAILED DESCRIPTION:
Records of women who had trophectoderm biopsy for sex selection over the last 3 years will be reviewed. Women will be divided into 3 groups: group 1 will comprise fertile women who had embryo biopsy for sex selection/family balancing, group 2 will comprise infertile women who had trophectoderm biopsy and group 3 will comprise infertile women who had IVF/ICSI without embryo biopsy.

The pregnancy and miscarriage rates of the groups will be compared. Before starting the embryo biopsy process couples were seen by a geneticist to assess the feasibility of the procedure for each couple. Couples were then counselled by a gynaecologist specialised in IVF to assess their fertility status and explain the whole procedure including the expected success rates and risks of IVF.

Women had standard pituitary down-regulation with GnRHa (Triptorelin 0.1mg, Decapeptyl® Ferring, Germany) day 7 after ovulation of previous cycle or on day 21 of the oral contraceptive cycles. GnRHa was continued for 2 weeks. Human menopausal gonadotrophin(HMG) (Merional ®IBSA) 150-300 IU/day was administered until the day of HCG administration, Transvaginal oocyte retrieval will be performed 34-36 h after the administration of HCG.

Day 5 embryos were incubated in calcium/Magnesium free culture. A laser beam was used to produce a hole in the zona pellucida. Trophectoderm cells were collected by gentle suction using the biopsy pipette.

Florescent in situ hybridization of the trophectoderm nuclei with probes specific to the X- and Y-chromosomes was performed. the embryos were frozen and the cycles deferred.The embryos were thawed in the following cycle and if possible 2 embryos of the desired sex were transferred.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF/ICSI

Exclusion Criteria:

* Women with expected poor ovarian response according to the Bologna criteria.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women who had IVF/ICSI over the past 3 years in Dar AlTeb subfertility centre will be included in the study
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | 5 weeks after embryo transfer
  presence of a gestational sac in vaginal ultrasound

SECONDARY OUTCOMES:
Miscarriage | 24 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Dar AlTeb subfertility centre, Giza, Egypt

REFERENCES:
- [Background] Greco E, Biricik A, Cotarelo RP, Iammarone E, Rubino P, Tesarik J, Fiorentino F, Minasi MG. Successful implantation and live birth of a healthy boy after triple biopsy and double vitrification of oocyte-embryo-blastocyst. Springerplus. 2015 Jan 14;4:22. doi: 10.1186/s40064-015-0788-y. eCollection 2015. PMID 25625041
- [Background] Rubino P, Cotarelo RP, Alteri A, Rega E, Vigano P, Giannini P. Trophectoderm biopsy performed by a double laser zona drilling: first safety evidence. Eur J Obstet Gynecol Reprod Biol. 2014 Oct;181:344-5. doi: 10.1016/j.ejogrb.2014.08.019. Epub 2014 Aug 27. No abstract available. PMID 25199461